CLINICAL TRIAL: NCT02496780
Title: The Impact of Insulin Therapy on Protein Turnover in Pre-Diabetic Cystic Fibrosis Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEDS-2015-23490
Record Dates: First submitted 2015-06-18; First posted 2015-07-14 (Estimated); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Insulin Aspart; Insulin Detemir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator): once or 3x daily injectable placebo (insulin diluent)
  Interventions: Drug: placebo
- basal insulin levemir (Experimental): once daily basal insulin therapy with insulin levemir
  Interventions: Drug: levemir insulin
- rapid-acting insulin Novolog (Experimental): pre-meal rapid-acting insulin 3x/day with insulin novolog
  Interventions: Drug: novolog insulin
- Healthy controls (No Intervention): Healthy controls matched by age, gender and BMI to CF participants. These participants are only used for baseline information, no intervention or outcome measure collected

INTERVENTIONS:
Drug: novolog insulin — 3x daily rapid-acting insulin
  Other Names: apart
  Arms: rapid-acting insulin Novolog
Drug: levemir insulin — basal insulin once a day
  Other Names: detemir
  Arms: basal insulin levemir
Drug: placebo — once or 3x daily
  Other Names: insulin diluent
  Arms: placebo

SUMMARY:
Insulin replacement therapy may be effective in breaking the cycle of protein catabolism, undernutrition and overall clinical deterioration in pre-diabetic, insulin insufficient CF youth because of its potent anabolic effect. A significant number of CF patients might benefit from this therapeutic approach with a substantial impact on morbidity and mortality.

DETAILED DESCRIPTION:
Insulin insufficiency related to pancreatic fibrosis and β-cell dysfunction is present in almost every cystic fibrosis (CF) patient. Progressive abnormalities in insulin secretion begin in childhood, and, in adults, CF related diabetes (CFRD) is eventually present in more than half of the CF population. CFRD is associated with weight loss, protein catabolism, loss of lean body mass (LBM), and early death from lung disease and malnutrition. The negative consequences of diabetes are just the "tip of the iceberg", since clinical deterioration has been documented to begin in the pre-diabetic period. Non-diabetic glucose tolerance abnormalities in CF are associated with protein catabolism, weight loss and lung function decline, all of which correlate with the severity of insulin secretory defects, suggesting a key pathologic role for insulin insufficiency. Insulin is a potent anabolic hormone, critical for maintenance of body weight and muscle mass. In a placebo-controlled clinical trial, insulin therapy improved body mass index (BMI) and LBM in patients with very early CFRD (CFRD without fasting hyperglycemia), and this is now standard care for these patients. There is growing preliminary evidence that insulin therapy is beneficial even earlier, in CF patients with pre-diabetes due to insulin insufficiency. Given the universal prevalence of insulin insufficiency in CF, the high lifetime risk of developing diabetes, the clinical impact of insulin insufficiency on protein catabolism and survival in CF, and the critical importance of maintaining body weight and LBM in this population, there is an urgent need to determine whether insulin replacement therapy should be instituted for anabolic purposes prior to the actual onset of diabetes and, if so, to ascertain the optimal regimen. The current protocol describes a double-blind, placebo-controlled trial to determine whether insulin therapy improves protein catabolism in youth with CF and abnormal glucose tolerance, and to explore differences in efficacy between multiple daily pre-meal insulin dosing (as is currently standard for early CFRD) versus a more convenient once daily basal insulin dose (as has been used in small uncontrolled pilot studies). The findings of this study will provide a mechanistic rationale for instituting insulin in youth with CF and pre-diabetes, and will inform both research studies and clinical practice as to the best regimen for insulin delivery in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cystic fibrosis, age 10-25 years
2. A standard routine annual OGTT performed within 12 months of randomization
3. Abnormal glucose tolerance, with a fasting glucose level <126 mg/dl and

   * The 1-hr OGTT glucose is ≥200 mg/dl but the 2-hr glucose is <140 (INDET), OR
   * The 2-hour OGTT glucose is 140-199 mg/dl (impaired glucose tolerance, IGT).

Exclusion Criteria:

1. Diagnosis of CFRD, Consensus Conference definition (45)
2. Previous organ transplant, or transplant imminent during study period
3. BMI percentile >95
4. Treatment with systemic glucocorticoids (nasal or inhaled glucocorticoids are acceptable)
5. Therapy with growth hormone or Megace
6. Nighttime continuous drip gastrostomy/jejunostomy feedings
7. Pregnancy or breast-feeding or plans to become pregnant during study period
8. Any change in medications during the 3 months prior to the study

   • Exception: the new corrector/potentiator combination drug lumacaftor/ivacaftor is expected to get FDA approval in early 2015, and most CF patients with severe genotypes, including many eligible for this proposal, will receive this drug. This is not a contraindication to participation in the current proposal (and participation in other studies is not contraindicated in the PROSPECT post-marketing drug study). Though the primary effects of the combination therapy appear to be apparent after 1 month, we will wait 6 months after initiation of lumacaftor/ivacaftor before enrollment in this study to make sure subjects are in a steady state.
9. Any anticipated change in medication during the 3 month study period
10. Acute illness in the 6 weeks prior to enrollment

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Moran, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
No, individual data will remain with the PI.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Basal Insulin Levemir | Rapid-acting Insulin Novolog | Healthy Controls
Started | 12 | 13 | 15 | 25
Completed | 11 | 9 | 10 | 20
Not Completed | 1 | 4 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Basal Insulin Levemir | Rapid-acting Insulin Novolog | Healthy Controls | Total
Number analyzed (Participants) | 11 | 11 | 15 | 20 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 6 | 10 | 25
  Between 18 and 65 years | 7 | 6 | 9 | 10 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 7 | 9 | 26
  Male | 7 | 5 | 8 | 11 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 11 | 10 | 13 | 18 | 52
  More than one race | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Endogenous Protein Breakdown (Flux) After 4 Weeks of Insulin/Placebo Therapy, CF Patients
Description: Primary endpoint. Determined from a stable isotope-labelled test meal. In the primary analysis, patients on both forms of insulin were first combined and compared to CF patients on placebo. In a second analysis, the two insulin types were separately compared to eachother and to placebo.
  Change in rate of endogenous protein breakdown (Ra-end) change from baseline (pre-treatment) and after 4 wks of study drug
Time Frame: 4 weeks
Population: Healthy controls did not participant in the primary aim
Measure: Mean (Standard Error); unit: µmol/kg(LBM)/min
Arm/Group | Placebo | Basal Insulin Levemir | Rapid-acting Insulin Novolog
Number analyzed (Participants) | 11 | 9 | 10
µmol/kg(LBM)/min | -0.01 (0.047) | 0.022 (0.046) | 0.0004 (0.06)

2. Secondary Outcome: Baseline Protein Turnover (Flux), CF Patients vs Healthy Controls
Description: Endogenous protein breakdown at baseline (Ra-end). CF patients vs healthy controls.
  Rate of endogenous protein breakdown (Ra-end), nadir (µmol/kg(LBM)/min)
Time Frame: baseline
Population: Note that for this secondary endpoint we assessed the baseline data of the entire CF population versus controls. Thus, in this pre-treatment population, all CF patients were included as a group regardless of what arm they were later randomized to. This was the only comparison between CF and healthy controls, who were matched for age, gender and BMI to CF participants.
Measure: Mean (Standard Error); unit: µmol/kg(LBM)/min
Groups:
- CF Total: all participants with CF
Arm/Group | CF Total | Healthy Controls
Number analyzed (Participants) | 37 | 20
µmol/kg(LBM)/min | 0.963 (0.135) | 0.921 (0.219)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 8 weeks. The subjects had their baseline test meal at time 0, insulin / placebo was given weeks 2-8, and the second test meal (for calculation of primary endpoint) was at 6 weeks.
Arm/Group | Placebo | Basal Insulin Levemir | Rapid-acting Insulin Novolog | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/15 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/15 | 0/25
Other Adverse Events (participants affected / at risk) | 2/12 | 4/13 | 4/15 | 5/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Basal Insulin Levemir (N=13) | Rapid-acting Insulin Novolog (N=15) | Healthy Controls (N=25)
unable to consume test meal (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
vomiting with test meal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CF pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
meal technical problems (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
hyperglycemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
covid center closure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
patient withdrawal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated before reaching the planned sample size, after a futility analysis suggested a full sample size would not lead to a positive result.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT02496780/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT02496780/ICF_001.pdf